CLINICAL TRIAL: NCT02620046
Title: A Phase 3b Open-label Study to Determine the Long-term Safety and Efficacy of Vedolizumab Subcutaneous in Subjects With Ulcerative Colitis and Crohn's Disease
Brief Title: A Study of Long-term Effects of Vedolizumab Subcutaneous in Adults With Ulcerative Colitis and Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN0002SC-3030; U1111-1168-0921 (Registry Identifier: WHO); 2015-000482-31 (EudraCT Number); JapicCTI-163220 (Registry Identifier: JapicCTI); MLN0002SC-3030CTIL (Registry Identifier: Israel); 16/LO/0110 (Registry Identifier: NRES); NL55765.056.16 (Registry Identifier: CCMO); 189751 (Registry Identifier: HC-CTD); 163300410A0052 (Registry Identifier: NREC); MOH_2017-01-05_000040 (Other: CRS)
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Colitis, Ulcerative; Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ulcerative Colitis: Vedolizumab 108 mg (Experimental): Participants with ulcerative colitis (UC) who completed the Maintenance Phase in MLN0002SC-3027 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3027 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3027 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
  Interventions: Drug: Vedolizumab SC
- Crohn's Disease: Vedolizumab 108 mg (Experimental): Participants with Crohn's disease (CD) who completed the Maintenance Phase in MLN0002SC-3031 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3031 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3031 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
  Interventions: Drug: Vedolizumab SC

INTERVENTIONS:
Drug: Vedolizumab SC — Vedolizumab SC 108 mg injection

SUMMARY:
The main aim of the study is to check for long-term side effects of Vedolizumab Subcutaneous (also known as Vedolizumab SC) in people with ulcerative colitis (UC) and Crohn's disease (CD). Vedolizumab SC will be given as an injection just under the skin. This type of injection is called a subcutaneous injection or SC for short. Another aim of the study is to collect information on whether the participant's condition remains under control or improves during and after treatment with Vedolizumab SC.

Participants who previously took part in studies MLN0002SC-3027 or MLN0002SC-3031 will be invited to visit the study clinic. At this visit, the study doctor will check if each participant can take part in this study.

For those who can take part, participants will receive a subcutaneous injection of vedolizumab SC either once a week or once every 2 weeks. How often each participant receives vedolizumab SC will depend on their results from the previous study and on how active their condition is. Participants might be able to self-inject vedolizumab SC after being trained by the study doctors. During this study, the dose of vedolizumab SC might be increased for participants whose condition worsens.

Participants will continue treatment with vedolizumab SC until it is approved in their particular country, the participant decides to stop treatment, or the sponsor stops the study. If the sponsor stops the study before vedolizumab SC is approved in all countries, the sponsor will make sure all affected participants will have access to vedolizumab SC outside of the study.

After their final dose of vedolizumab SC, participants will visit the clinic 18 weeks later for a final check-up. Then, the clinic will telephone the participants 6 months after their final dose of vedolizumab SC to check if they have any health problems.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab subcutaneous (vedolizumab SC). Vedolizumab SC is being tested to assess its long-term safety and effectiveness in treating participants with UC or CD. This study will look at the long-term side effects and response/remission of UC and CD in participants who received vedolizumab SC in a prior vedolizumab SC study.

The study will enroll up to 692 patients. All participants enrolled in this study will have previously participated in the MLN0002SC-3027 or MLN0002SC-3031 study. Participants who completed the Maintenance Period (Week 52) in their previous study, or who did not achieve a clinical response at Week 6 but who did achieve a clinical response at Week 14 after having received a third vedolizumab IV infusion at Week 6 in their previous study, will receive open-label vedolizumab SC 108 mg, once every 2 weeks (Q2W). Participants who withdrew early from the Maintenance Period of their previous study due to disease worsening or need for rescue medications will receive open-label vedolizumab SC 108 mg, once every week (QW). Participants receiving SC 108 mg Q2W who experience treatment failure (disease worsening or need for rescue medications while in the current study will be dose escalated to vedolizumab SC 108 mg QW.

This multi-center trial will be conducted worldwide. Participation in this vedolizumab SC study will continue until vedolizumab SC becomes commercially available, the participant withdraws from the study, or the sponsor decides to close the study. Participants will make multiple visits to the clinic, plus a final visit 18 weeks after last dose of study drug for a follow-up assessment. Participants will also participate in a long-term safety follow-up, by phone, at 6 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Prior participation in Study MLN0002SC-3027 or MLN0002SC-3031, and, in the opinion of the investigator, tolerated the study drug well. Early withdrawal from Study MLN0002SC-3027 or MLN0002SC-3031 must have been due to treatment failure during the Maintenance Period.

Exclusion Criteria:

1. Surgical intervention for IBD during or after participation in Study MLN0002SC-3027 or MLN0002SC-3031, or at any time during this study.
2. Chronic or severe infection, or, any new, unstable, or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, neurologic, oncologic, or other medical disorder developed during or after participation in a prior vedolizumab study that, in the opinion of the investigator, would confound the study results or compromise participant safety.
3. Withdrawal from Study MLN0002SC-3027 or MLN0002SC-3031 due to a study-drug related adverse event (AE).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (301):
- United States (47):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Rocky Mountain Clinical Research, LLC, Wheat Ridge, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Middlesex Gastroenterology Associates, Middletown, Connecticut
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - L & L Research Choices, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - BRCR Medical Center, Inc., Pembroke Pines, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Grand Teton Research Group, PLL, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Research Concierge, LLC, Owensboro, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Long Island Clinical Research Associates, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Gastro-Enterology Research of Lima, Lima, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Main Line Gastroenterology Associates, Perkasie, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Gastroenterology, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Virginia Mason Seattle Main Clinic, Seattle, Washington
  - Allegiance Research Specialists, LLC, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro Medico Viamonte SRL, Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (14):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Tennyson Centre Day Hospital, Kurralta Park, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Monash Medical Centre Clayton, Bentleigh East, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (7):
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint-Lucas, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Kennedylaan, Kortrijk
  - ZNA Jan Palfijn, Merksem
  - Clinique Saint-Pierre, Ottignies
  - AZ Delta, Roeselare
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
- Brazil (9):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - HUGG - Hospital Universitario Gaffree e Guinle, Rio de Janeiro, Rio Do Janeiro
  - HUCFF-UFRJ - Hospital Universitario Clementino Fraga Filho - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio Do Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Irmandade da Santa Casa da Misericordia de Santos, Santos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
- Bulgaria (14):
  - "MHAT Avis - Medica" OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - MHAT - Silistra AD, Silistra
  - MC "Tsaritsa Yoanna' EOOD, Sliven
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - Second MHAT - Sofia AD, Sofia
  - "City Clinic UMHAC" EOOD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - UMHAT 'Sveta Anna' AD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Canada (5):
  - Zeidler Ledcor Centre - University of Alberta, Edmonton, Alberta
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
- Croatia (5):
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Special Hospital Medico, Rijeka
  - Clinical Hospital Dubrava, Zagreb
  - University hospital centre Zagreb, Zagreb
- Czechia (7):
  - CCBR - Czech Brno, s.r.o.., Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - A-SHINE s.r.o., Pilsen
  - CLINTRIAL s.r.o., Prague
  - CCBR Czech Prague, s.r.o., Prague
  - Axon Clinical s.r.o., Prague
  - Nemocnice Tabor a.s., Tábor
- Denmark (2):
  - Odense Universitetshospital, Odense C
  - Regionshospitalet Silkeborg, Silkeborg
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Germany (12):
  - LMU - Campus Grosshadern, Munich, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - EUGASTRO GmbH, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - Charite - Campus Virchow-Klinikum, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
- Hungary (12):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - Pecsi Tudomanyegyetem, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (10):
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (27):
  - Yokoyama IBD Clinic, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Tokushukai Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Hamamatsu South Hospital, Hamamatsu, Shizuoka
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City, Tokyo-To
  - Jikei University Hospital, Minatoku, Tokyo-To
  - Kitasato University Kitasato Institute Hospital, Minatoku, Tokyo-To
  - Kyorin University Hospital, Mitaka-shi, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo-To
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Republican Hospital, Public Institution, Klaipėda
  - Klaipeda University Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius
- Mexico (7):
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Centro de Investigacion Farmacologica del Bajio, S.C., León, Guanajuato
  - iBiomed Guadalajara, Zapopan, Jalisco
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Christus Muguerza Sur S.A. de C.V., Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (14):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - NZOZ Vitamed, Bydgoszcz
  - SP CSK im. prof. K. Gibinskiego SUM, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - SPZOZ Uniwersytecki Szpital Klin. nr 1 im.N.Barlickiego UM, Lodz
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - GASTROMED Sp. z o.o., Lublin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
- Romania (3):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Russia (10):
  - Kazan State Medical University, Kazan'
  - TSBIH "Territorial Clinical Hospital", Krasnoyarsk
  - FSBIH "Central Clinical Hospital of Russian Academy of Sciences", Moscow
  - LLC "Novosibirsk GastroCenter", Novosibirsk
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - SBEI HPE "Rostov State Medical University" of the MoH of the RF, Rostov-on-Don
  - SPb SBIH "City Hospital of Saint Martyr Elizaveta", Saint Petersburg
  - LLC "RIAT SPb", Saint Petersburg
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
- Serbia (8):
  - Clinical Center of Serbia, Belgrade
  - Clinical Helth Centre Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Gastroped s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
- South Africa (3):
  - Dr CCM Ziady Practice, Pretoria, Gauteng
  - Dr MJ Prins Practice, Cape Town, Western Cape
  - Dr JP Wright Practice, Cape Town, Western Cape
- South Korea (8):
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
- Sweden (2):
  - Karolinska Universitetssjukhuset - Solna, Stockholm
  - Danderyds Sjukhus, Stockholm
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Ankara University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
  - Kocaeli Derince Training and Research Hospital, Kocaeli
  - Mersin University Medical Faculty, Mersin
- Ukraine (15):
  - RCNECRCH Dept of Surgery, SHEI Ukr BSMU, Chernivtsi
  - SI Institute of Gastroenterology of NAMSU Dept of Stomach & Duodenum Diseases, D&ThN SI DMA of MoHU, Dnipro
  - Regional CH Dep of Gastroenterology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - CI A.and O. Tropiny City Clinical Hospital, Kherson
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv
  - MI of Healthcare Kyiv RCH P.L. Shupyk NMA of PGE, Kyiv
  - Kyiv CCH #12 Dept of Therapy O.O.Bogomolets NMU, Kyiv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - CI Odesa Regional Clinical Hospital, Odesa
  - Ternopil University Hospital, Ternopil
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia RCH of Veterans of War Dept of Therapy#1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - CI City Hospital #1, Zaporizhzhia
- United Kingdom (8):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Whipps Cross University Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - St George's Hospital, London, Greater London
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - University Hospital Coventry, Coventry, West Midlands
  - Royal Wolverhampton hospital, Wolverhampton, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ungaro RC, Kadali H, Zhang W, Adsul S, Reinisch W. Impact of Concomitant 5-Aminosalicylic Acid Therapy on Vedolizumab Efficacy and Safety in Inflammatory Bowel Disease: Post Hoc Analyses of Clinical Trial Data. J Crohns Colitis. 2023 Dec 30;17(12):1949-1961. doi: 10.1093/ecco-jcc/jjad113. PMID 37492976
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60274db2bf003ab498d5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 15 April 2016 to 12 June 2024.
Pre-assignment Details: Participants who had previously participated in Study MLN0002SC-3027 [NCT02611830] or MLN0002SC-3031 [NCT02611817] and were eligible to participate received vedolizumab subcutaneously (SC) [either 108 milligrams (mg) once every two weeks (Q2W) or once per week (QW)] in the disease groups of Ulcerative Colitis and Crohn's Disease in this study. Data is presented accordingly.
Groups:
- Ulcerative Colitis: Vedolizumab 108 mg: Participants with ulcerative colitis (UC) who completed the Maintenance Phase in MLN0002SC-3027 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3027 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas participants who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3027 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
- Crohn's Disease: Vedolizumab 108 mg: Participants with Crohn's disease (CD) who completed the Maintenance Phase in MLN0002SC-3031 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3031 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas participants who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3031 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
Period: Overall Study
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg | Crohn's Disease: Vedolizumab 108 mg
Started | 288 | 458
Completed | 125 | 162
Not Completed | 163 | 296
Not completed — Adverse Event | 22 | 42
Not completed — Lost to Follow-up | 4 | 10
Not completed — Withdrawal by Subject | 36 | 66
Not completed — Site Termination | 3 | 3
Not completed — Pregnancy | 3 | 7
Not completed — Lack of Efficacy | 81 | 146
Not completed — Leukopenia or Lymphopenia | 1 | 0
Not completed — Reason Not Specified | 13 | 21
Not completed — Significant Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) included all participants who had received at least 1 dose of study medication in this study (MLN0002SC-3030). As per planned analysis, baseline characteristics data was collected and presented per disease condition in the arm groups, 'Ulcerative Colitis: Vedolizumab 108 mg' and 'Crohn's Disease: Vedolizumab 108 mg'.
Groups:
- Ulcerative Colitis: Vedolizumab 108 mg: Participants with UC who completed the Maintenance Phase in MLN0002SC-3027 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3027 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas participants who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3027 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
- Crohn's Disease: Vedolizumab 108 mg: Participants with CD who completed the Maintenance Phase in MLN0002SC-3031 (Week 52 assessment) or who did not achieve a clinical response at Week 6 in MLN0002SC-3031 but who did achieve a clinical response at Week 14 of the parent study after having received a third vedolizumab IV infusion at Week 6 in the parent study received vedolizumab SC 108 mg Q2W in this study whereas participants who withdrew early from the Maintenance Phase (at Week 14 onwards) in MLN0002SC-3031 due to disease worsening or need for rescue medications received vedolizumab SC 108 mg QW.
- Total: Total of all reporting groups
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg | Crohn's Disease: Vedolizumab 108 mg | Total
Number analyzed (Participants) | 288 | 458 | 746
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 265 | 440 | 705
  >=65 years | 23 | 18 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 214 | 334
  Male | 168 | 244 | 412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 34 | 94 | 128
  Unknown or Not Reported | 253 | 361 | 614
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 58 | 28 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 9 | 11
  White | 226 | 417 | 643
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs Adjusted by Duration of Participant's Exposure to Long-term Vedolizumab Treatment
Description: A TEAE was defined as an adverse event (AE) that started or worsened on or after study Day 1 (defined as day first dosed) and no more than 18 weeks after the last dose of study drug. An SAE was defined as any untoward medical occurrence that occurs at any dose and resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was an important medical event such as acute liver failure, pulmonary hypertension, or confirmed or suspected transmission of an infectious agent by a medicinal product. Participant years is defined as the total exposure-time of the participants in the respective treatment group. Incidence per 100 participant years is defined as (Number of participants with events*100/participant years). As per planned analysis, data for this outcome measure is grouped and presented per disease condition.
Time Frame: Up to 97.9 months
Population: The SAF included all participants who had received at least 1 dose of study medication during this study (MLN0002SC-3030).
Measure: Number; unit: events per 100 participant years
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg | Crohn's Disease: Vedolizumab 108 mg
Number analyzed (Participants) | 288 | 458
events per 100 participant years
  TEAEs | 22.9 | 28.0
  Serious TEAEs | 6.5 | 8.7

2. Secondary Outcome: Number of Adverse Events of Special Interest (AESIs) Adjusted by Duration of Participant's Exposure to Long-term Vedolizumab Treatment
Description: AESIs included hypersensitivity reactions (including injections site reactions), serious infections, malignancies, hepatotoxicity (abnormal liver function test) and progressive multifocal leukoencephalopathy (PML). Participant years is defined as the total exposure-time of the participants in the respective treatment group. Incidence per 100 participant years is defined as (Number of participants with events*100/participant years). As per planned analysis, data for this outcome measure is grouped and presented per disease condition.
Time Frame: Up to 97.9 months
Population: as for outcome 1
Measure: Number; unit: events per 100 participant years
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg | Crohn's Disease: Vedolizumab 108 mg
Number analyzed (Participants) | 288 | 458
events per 100 participant years | 16.3 | 17.4

3. Secondary Outcome: Number of Participants With Ulcerative Colitis Achieving Partial Mayo Scoring Clinical Response at Week 48
Description: Clinical response is defined as a decrease in the partial Mayo score of at least 2 points and ≥25% from baseline, with an accompanying decrease in rectal bleeding subscore of ≥1 point from baseline or absolute rectal bleeding subscore of ≤1 point. As per planned analysis, data for this outcome measure is grouped and presented for participants with ulcerative colitis.
Time Frame: Week 48
Population: Full Analysis Set (FAS) included all enrolled participants of this study MLN0002SC-3030. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg
Number analyzed (Participants) | 288
Participants | 168

4. Secondary Outcome: Number of Participants With Crohn's Disease Achieving Clinical Response Based on Harvey-Bradshaw Index (HBI) Scores at Week 48
Description: Clinical response is defined as a decrease in HBI score of ≥3 points from baseline in CD participants (randomized early terminator CD participants only [defined as randomized CD participants withdrawn from the parent study between Week 6 and Week 52]). As per planned analysis, data for this outcome measure is grouped and presented for participants with Crohn's disease.
Time Frame: Week 48
Population: FAS included all enrolled participants of this study MLN0002SC-3030. Overall number analyzed is the number of randomized CD participants withdrawn from the parent study between Week 6 and Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease: Vedolizumab 108 mg
Number analyzed (Participants) | 114
Participants | 32

5. Secondary Outcome: Number of Participants With Ulcerative Colitis Achieving Clinical Remission Based on Partial Mayo Score
Description: Clinical remission is defined as a partial Mayo score of ≤2 with no individual subscore >1. As per planned analysis, data for this outcome measure is grouped and presented for participants with ulcerative colitis.
Time Frame: Week 48
Population: FAS included all enrolled participants of this study MLN0002SC-3030.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulcerative Colitis: Vedolizumab 108 mg
Number analyzed (Participants) | 288
Participants | 150

6. Secondary Outcome: Number of Participants With Crohn's Disease Achieving Clinical Remission Based on Harvey-Bradshaw Index (HBI) Scores
Description: Clinical remission is defined as total HBI score of ≤4 points. As per planned analysis, data for this outcome measure is grouped and presented for participants with Crohn's disease.
Time Frame: Week 48
Population: FAS included all enrolled participants of this study MLN0002SC-3030.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease: Vedolizumab 108 mg
Number analyzed (Participants) | 458
Participants | 217

ADVERSE EVENTS:
Time Frame: Up to 97.9 months
Description: The SAF included all participants who had received at least 1 dose of study medication in this study (MLN0002SC-3030). Adverse events and All-cause mortality are presented as per the dosing regimen.
Groups:
- Ulcerative Colitis: Only Vedolizumab Q2W: Participants with UC who received vedolizumab SC 108 mg Q2W in this study were included in this arm group.
- Ulcerative Colitis: Only Vedolizumab QW: Participants with UC who received vedolizumab SC 108 mg QW in this study were included in this arm group.
- Ulcerative Colitis: Vedolizumab Dose Escalation From Q2W to QW: Participants with UC who experienced treatment failure (i.e., disease worsening or need for rescue medications) while receiving vedolizumab 108 mg Q2W during this study and underwent dose escalation to receive vedolizumab SC 108 mg QW were included in this arm group.
- Crohn's Disease: Only Vedolizumab Q2W: Participants with CD who received vedolizumab SC 108 mg Q2W in this study were included in this arm group.
- Crohn's Disease: Only Vedolizumab QW: Participants with CD who received vedolizumab SC 108 mg QW in this study were included in this arm group.
- Crohn's Disease: Vedolizumab Dose Escalation From Q2W to QW: Participants with CD who experienced treatment failure (i.e., disease worsening or need for rescue medications) while receiving vedolizumab 108 mg Q2W during this study and underwent dose escalation to receive vedolizumab SC 108 mg QW were included in this arm group.
Arm/Group | Ulcerative Colitis: Only Vedolizumab Q2W | Ulcerative Colitis: Only Vedolizumab QW | Ulcerative Colitis: Vedolizumab Dose Escalation From Q2W to QW | Crohn's Disease: Only Vedolizumab Q2W | Crohn's Disease: Only Vedolizumab QW | Crohn's Disease: Vedolizumab Dose Escalation From Q2W to QW
All-Cause Mortality (participants affected / at risk) | 3/163 | 0/60 | 0/65 | 2/239 | 0/117 | 0/102
Serious Adverse Events (participants affected / at risk) | 29/163 | 12/60 | 24/65 | 55/239 | 35/117 | 31/102
Other Adverse Events (participants affected / at risk) | 94/163 | 41/60 | 55/65 | 151/239 | 78/117 | 90/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ulcerative Colitis: Only Vedolizumab Q2W (N=163) | Ulcerative Colitis: Only Vedolizumab QW (N=60) | Ulcerative Colitis: Vedolizumab Dose Escalation From Q2W to QW (N=65) | Crohn's Disease: Only Vedolizumab Q2W (N=239) | Crohn's Disease: Only Vedolizumab QW (N=117) | Crohn's Disease: Vedolizumab Dose Escalation From Q2W to QW (N=102)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 6 | 3 | 3 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 4 | 7 | 11 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 10 | 14
Cytomegalovirus enteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0/61 | 0/27 | 0/32 | 1/106 | 0/63 | 0/45 — Number of participants at risk in each arm is based on the female population in this study.
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal organ contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Ileal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/61 | 0/27 | 0/32 | 1/106 | 0/63 | 0/45 — Number of participants at risk in each arm is based on the female population in this study.
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal fibrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Liver contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/102 | 0/33 | 0/33 | 1/133 | 0/54 | 0/57 — Number of participants at risk in each arm is based on the male population in this study.
Prostatitis (Reproductive system and breast disorders) | 0/102 | 0/33 | 0/33 | 1/133 | 0/54 | 0/57 — Number of participants at risk in each arm is based on the male population in this study.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary pneumatocele (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/102 | 0/33 | 0/33 | 1/133 | 0/54 | 0/57 — Number of participants at risk in each arm is based on the male population in this study.
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/61 | 0/27 | 0/32 | 0/106 | 0/63 | 1/45 — Number of participants at risk in each arm is based on the female population in this study.
Vascular headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ulcerative Colitis: Only Vedolizumab Q2W (N=163) | Ulcerative Colitis: Only Vedolizumab QW (N=60) | Ulcerative Colitis: Vedolizumab Dose Escalation From Q2W to QW (N=65) | Crohn's Disease: Only Vedolizumab Q2W (N=239) | Crohn's Disease: Only Vedolizumab QW (N=117) | Crohn's Disease: Vedolizumab Dose Escalation From Q2W to QW (N=102)
Abdominal pain (Gastrointestinal disorders) | 8 | 3 | 2 | 33 | 20 | 15
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 10 | 3 | 7
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 9 | 14 | 3 | 6
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 5 | 34 | 14 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 3 | 14 | 4 | 9
Blood creatine phosphokinase increased (Investigations) | 8 | 4 | 4 | 13 | 2 | 5
Bronchitis (Infections and infestations) | 9 | 1 | 6 | 16 | 8 | 8
COVID-19 (Infections and infestations) | 24 | 2 | 5 | 29 | 4 | 9
Colitis ulcerative (Gastrointestinal disorders) | 8 | 14 | 33 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 4 | 10 | 2 | 8
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 26 | 30 | 53
Diarrhoea (Gastrointestinal disorders) | 12 | 2 | 8 | 18 | 12 | 10
Fatigue (General disorders) | 6 | 0 | 1 | 13 | 5 | 5
Gastroenteritis (Infections and infestations) | 4 | 4 | 2 | 11 | 6 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 0 | 6
Headache (Nervous system disorders) | 8 | 3 | 7 | 19 | 5 | 14
Herpes zoster (Infections and infestations) | 4 | 1 | 4 | 2 | 5 | 1
Hypertension (Vascular disorders) | 8 | 0 | 4 | 12 | 3 | 5
Influenza (Infections and infestations) | 4 | 3 | 7 | 12 | 5 | 3
Injection site erythema (General disorders) | 2 | 5 | 1 | 3 | 2 | 1
Injection site reaction (General disorders) | 2 | 4 | 0 | 2 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 3 | 1 | 3
Nasopharyngitis (Infections and infestations) | 23 | 11 | 15 | 26 | 16 | 20
Nausea (Gastrointestinal disorders) | 7 | 1 | 3 | 14 | 7 | 13
Pharyngitis (Infections and infestations) | 7 | 1 | 4 | 6 | 6 | 3
Pneumonia (Infections and infestations) | 3 | 1 | 4 | 3 | 1 | 2
Pyrexia (General disorders) | 5 | 4 | 3 | 12 | 9 | 10
Sinusitis (Infections and infestations) | 9 | 2 | 4 | 12 | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 28 | 6 | 7 | 38 | 13 | 18
Urinary tract infection (Infections and infestations) | 8 | 2 | 1 | 12 | 5 | 9
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2 | 13 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02620046/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02620046/SAP_001.pdf